CLINICAL TRIAL: NCT05197114
Title: Assessing the Feasibility and Acceptability of a Virtual Food Skills Program for Children With Type 1 Diabetes During COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Vanita Pais, Registered Dietitian, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1000076894
Record Dates: First submitted 2021-12-29; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): There will be one arm to the study, and all participants will be receiving the intervention.
  Interventions: Other: summerlunch+ At Home Food Skills Program

INTERVENTIONS:
Other: summerlunch+ At Home Food Skills Program — The summerlunch+ At Home program a virtual eight-week food skills program that teaches cooking, nutrition and environmental sustainability to children. The program has been adapted for those with Type 1 Diabetes to teach important food skills specific to diabetes management.

SUMMARY:
Food forms an integral part of diabetes management. As children mature into young adults, they must learn to adopt lifestyle behaviours critical for optimal diabetes care. The development of food preparation and cooking skills at a young age may help to facilitate healthy food choices in children and provide a solid foundation for young adulthood. Food skills workshops are effective interventions that have been shown to improve food literacy and healthy eating in the general pediatric population. However, food skills programs have not been adequately evaluated in children with type 1 diabetes. Further, virtual programs are not well assessed, which can increase the accessibility of food education during the pandemic and in the future.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for over one year

Exclusion Criteria:

* Type 1 diabetes for less than one year, non-English speaking, do not have access to a computer or internet

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-01-25 (Estimated); Primary Completion 2022-03-25 (Estimated); Study Completion 2022-09-25 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability of the virtual summerlunch+At Home program | Two months
  Questionnaire
Feasibility and acceptability of the virtual summerlunch+At Home program | Three months
Feasibility and acceptability of the virtual summerlunch+At Home program | Six months
  Questionaire

SECONDARY OUTCOMES:
The impact of the program on food literacy skills children's attitude towards cooking, cooking confidence, food knowledge and food preferences - | Two months, three months and six months
  Questionnaire to measure the change in food literacy skills before and after the program.
Changes in glycemic control as measured through HbA1C levels | Two months, three months and six months
  Routine blood work

CONTACTS AND LOCATIONS:
Overall Officials: Vanita Pais, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No